CLINICAL TRIAL: NCT04469517
Title: Influence of Hypoxic Induced Factors in Patients With Hereditary Hemorrhagic Telangiectasia (HHT)
Brief Title: Influence of Hypoxic Induced Factors in Patients With Hereditary Hemorrhagic Telangiectasia
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Freya Droege, Principle Investigator, Speaker of Westgerman HHT Center, University Hospital, Essen
Other Study IDs: HIF in HHT
Record Dates: First submitted 2020-07-08; First posted 2020-07-14 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Hereditary Hemorrhagic Telangiectasia
Keywords: hereditary hemorrhagic telangiectasia
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HHT: patients with HHT
  Interventions: Other: hypoxic induced factors
- control: persons age- and sex matched who do not suffer from HHT nor their first or second degree relatives
  Interventions: Other: hypoxic induced factors

INTERVENTIONS:
Other: hypoxic induced factors — hypoxic induced factors analyzed in blood sample

SUMMARY:
Patients with hereditary hemorrhagic telangiectasia (HHT) suffer from an inherited disorder leading to systemic vascular malformations. Mutations in several genes of the transforming growth factor (TGF)-β superfamily pathway influence angiogenesis in patients with HHT. The genetic loss of ALK1 or ENG alone are not sufficient to induce AVMs; environmental insults that could trigger angiogenesis (e.g. wounding) are also needed. In this study it will be analyzed if hypoxic induced factors could have an influence on the disease HHT.

DETAILED DESCRIPTION:
Hereditary hemorrhagic telangiectasia (HHT) is characterized by systemic vascular malformations leading to recurrent bleedings and shunt formation especially in the liver, lungs and the brain. The underlying pathogenic HHT mechanism remains unclear. The wide variability in age of onset and severity of symptoms amongst patients, even within the same family, suggests several factors contribute to the complexity of this disease. Mutations in several genes of the transforming growth factor (TGF)-β superfamily pathway influence angiogenesis in patients with HHT. The genetic loss of ALK1 or ENG alone are not sufficient to induce AVMs; environmental insults that could trigger angiogenesis (e.g. wounding) are also needed. In this study it will be analyzed if hypoxic induced factors could have an influence on the disease HHT.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed HHT (genetic testing and/ or fulfill at least 3 Curacao Criteria)
* older than 17 years
* ability to consent

Exclusion Criteria:

* if inclusion Criteria are not met

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed hereditary hemorrhagic telangiectasie (HHT)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Differences in hypoxic induced factors | 12 months
  Differences in hypoxic induced factors analyzed in blood samples from patients with HHT and healthy controls

SECONDARY OUTCOMES:
Correlation of level of hypoxic induced factors and disease severity | 12 months
  Correlation of level of hypoxic induced factors in patients' blood sample and their disease severity

CONTACTS AND LOCATIONS:
Overall Officials: Freya Droege, MD, Principal Investigator — University hospital Essen Otorhinolaryngology, Hufelandstr. 55, 45147 Essen, Germany
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kjeldsen AD, Vase P, Green A. [Hereditary hemorrhagic telangiectasia. A population-based study on prevalence and mortality among Danish HHT patients]. Ugeskr Laeger. 2000 Jun 19;162(25):3597-601. Danish. PMID 11016284
- [Background] Shovlin CL, Guttmacher AE, Buscarini E, Faughnan ME, Hyland RH, Westermann CJ, Kjeldsen AD, Plauchu H. Diagnostic criteria for hereditary hemorrhagic telangiectasia (Rendu-Osler-Weber syndrome). Am J Med Genet. 2000 Mar 6;91(1):66-7. doi: 10.1002/(sici)1096-8628(20000306)91:13.0.co;2-p. PMID 10751092
- [Background] Sanchez-Elsner T, Botella LM, Velasco B, Corbi A, Attisano L, Bernabeu C. Synergistic cooperation between hypoxia and transforming growth factor-beta pathways on human vascular endothelial growth factor gene expression. J Biol Chem. 2001 Oct 19;276(42):38527-35. doi: 10.1074/jbc.M104536200. Epub 2001 Aug 2. PMID 11486006
- [Background] Park SO, Wankhede M, Lee YJ, Choi EJ, Fliess N, Choe SW, Oh SH, Walter G, Raizada MK, Sorg BS, Oh SP. Real-time imaging of de novo arteriovenous malformation in a mouse model of hereditary hemorrhagic telangiectasia. J Clin Invest. 2009 Nov;119(11):3487-96. doi: 10.1172/JCI39482. Epub 2009 Oct 1. PMID 19805914
- [Background] Attisano L, Wrana JL. Smads as transcriptional co-modulators. Curr Opin Cell Biol. 2000 Apr;12(2):235-43. doi: 10.1016/s0955-0674(99)00081-2. PMID 10712925